CLINICAL TRIAL: NCT02358915
Title: A Two-step Training Paradigm for Voluntary Control of the Peri-auricular Muscles
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Carolee Winstein, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-14-00672
Record Dates: First submitted 2015-01-29; First posted 2015-02-09 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Non-disabled Volunteers; Lacking Voluntary Control of Ear Muscles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peri-auricular muscles voluntary contraction training paradigm (Experimental): The whole training paradigm consists of two steps. At the first step of training, the electrical stimulation (FastStart neuromuscular electrical stimulator) will be applied to facilitate the voluntary contractions of the ear muscles, and the motion of the outer ear in two directions (up/down, forward/backward) will be videotaped and played back to the participants so that they can get real-time visual feedback about their ear movement. At the second step of training, surface EMG electrodes will be placed on the skin around participants' ears. During the training, they are required to move a cursor to a specific target that will randomly appear on the computer screen. The cursor will be controlled by the electrical signal from the contraction of their bilateral peri-auricular muscles. In the computer game, contraction of the left ear muscles will move the cursor to the left side and contraction of your right ear muscles will move the cursor to the right side.
  Interventions: Device: FastStart neuromuscular electrical stimulator

INTERVENTIONS:
Device: FastStart neuromuscular electrical stimulator
  Other Names: Biosemi Active two EMG measurement system

SUMMARY:
The current study intends to test the effectiveness of a two-step training paradigm for a set of skeletal muscles, which are above and behind the external portion of the ear (Peri-auricular muscles).

DETAILED DESCRIPTION:
Survivors of spinal cord injury (SCI) usually have severe mobility limitation due to their paralysis.In order to improve the independence of living for those patients, scientists and engineers invented many different types of assistive devices, such as breath controlled "sip and puff" devices, speech controlled devices, eye movement controlled devices, and head movement controlled devices. However, one limitation of the previous designs is that they all require usurping the intact function of a functional organ like mouth or eyes. A recent design by Reach Bionic's company takes advantage of a set of ear muscles-the peri-auricular muscles-that are present in more than 95% of the population, but do not serve any physiologic function in humans. These muscles are innervated by branches of cranial nerves that are controlled through the brain stem, above the spinal cord. Therefore, it is unlikely they will be affected even by a very high SCI. The design intention is to translate the ear contraction signal from the muscles into the meaningful control signal to direct a wheelchair or operate a computer cursor in a fashion to a joystick or mouse. However, since most people do not have the ability to voluntarily contract their ear muscles, the question remains how to best learn to contract our ear muscles and design an effective training paradigm.

Since norm volunteers will have the same voluntary control of their peri-auricular muscles as the patients suffering from spinal cord injury, thus, the investigators are going to test the effectiveness of our two-step training paradigm among the healthy participants at this explorative stage.

In specific, at the first step of training, participants will be asked to voluntarily contract their ear muscles with the facilitation of electrical stimulation. At the second step of training, they will take part in a computer game and will be asked to move a cursor to a specific target that will randomly appear on the computer screen. The cursor will be controlled by the electrical activities produced by the ear muscles contractions that will be captured by surface electromyography (EMG) signals.

The computer game performance of each participant before and after the second step of training with surface EMG signals feedback and the mean surface EMG signal amplitude of the auricular muscles at the maximum voluntary contraction at baseline, after the first step of training, and after the second step of training will be compared.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* can't control their peri-auricular muscles at the beginning of the study (no visible movement of the ears on command).

Exclusion Criteria:

* Suffering any comorbid neuromuscular disease.
* Having a history of severe traumatic brain injury.
* Demonstrating cognitive impairment that would prevent them from providing inform consent or following the directions of the study protocol.
* Having a history of migraine headaches that could be exacerbated with the use of the electrical stimulation or the prolonged training sessions.
* Temporomandibular Joint (TMJ) dysfunction that could lead to unusual discomfort following training session.
* Having a history of prior seizure.
* Being implanted with pacemaker or defibrillators.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
The surface EMG signal amplitude of the auricular muscles at the maximum voluntary contraction | Up to 5 weeks

SECONDARY OUTCOMES:
The computer game performance score | Up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolee J. Winstein, Ph.D, Principal Investigator — University of Southern California; Baker Lucinda, Ph.D, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California-Health Sciences Campus, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chanthaphun S, Heck SL, Winstein CJ, Baker L. Development of a training paradigm for voluntary control of the peri-auricular muscles: a feasibility study. J Neuroeng Rehabil. 2019 Jun 14;16(1):75. doi: 10.1186/s12984-019-0540-x. PMID 31200729